CLINICAL TRIAL: NCT03391362
Title: Stereotactic Radiation in Patients With Small Cell Lung Cancer and 1-10 Brain Metastases: A Single Arm, Phase II Trial
Brief Title: Stereotactic Radiation in Patients With Small Cell Lung Cancer and 1-10 Brain Metastases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ayal Aizer, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-550
Record Dates: First submitted 2017-12-21; First posted 2018-01-05 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Brain Metastases; Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Brain Metastases; Brain metastasis; Lung cancer; Stereotactic radiation; Stereotactic radiosurgery; SRS; Stereotactic; Radiation; Quality of life; Neurocognitive; Neurocognition
MeSH Terms: conditions — Brain Neoplasms; Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Radiation (Experimental): * Stereotactic radiation will begin within 14 days of the MRI used for radiation planning
  * Lesions <2 cm in maximum diameter will be treated with stereotactic radiosurgery, generally 20 Gy in 1 fraction
  * Lesions between 2.0 and 3.0 cm in maximum diameter will generally be treated to 18 Gy in 1 fraction
  * Lesions >3 cm will be generally be treated with stereotactic radiotherapy to 30 Gy in 5 fractions
  Interventions: Radiation: Stereotactic Radiation

INTERVENTIONS:
Radiation: Stereotactic Radiation — Stereotactic radiation involves using a high dose of radiation that only targets the specific metastases

SUMMARY:
This research study is studying stereotactic radiation (focused/pinpoint radiation that targets each individual tumor but not the surrounding brain) instead of whole-brain radiation (radiation targeting the entire brain) as a possible treatment for patients with small cell lung cancer and 1-10 brain metastases.

The intervention involved in this study is:

-Stereotactic (focused, pinpoint) radiation

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational treatment, in this case stereotactic radiation, to learn whether this treatment works in treating a specific disease. "Investigational" means that the treatment is being studied.

In patients with a limited number of brain metastases (spread of a cancer that started outside of the brain to the brain itself) the standard radiation option is stereotactic radiation, which involves using a high dose of radiation that only targets the specific metastases that are visible on imaging of the brain, not the whole brain itself. However, studies evaluating the role of stereotactic radiation to treat brain metastases generally excluded patients with small cell lung cancer. Therefore, among patients with small cell lung cancer and brain metastases, the typical treatment that has been offered is whole brain radiation. However, whole brain radiation has deleterious associated side effects including significant fatigue and permanent memory/attention problems. The investigators are studying whether stereotactic radiation can be effectively utilized for patients with small cell lung cancer and brain metastases in order to avoid such side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a biopsy-proven tumor consistent with small cell lung cancer and intracranial lesions radiographically consistent with or pathologically proven to be brain metastases. Patients who have undergone prior systemic therapy are eligible. Patients who have undergone resection of one or more brain metastases but who have not yet started adjuvant radiotherapy are eligible for the study.
* 1-10 definitive intracranial lesions must be present on MRI of the brain.
* Age >=18 years at diagnosis of brain metastases.

Exclusion Criteria:

* Participants who have undergone prior radiation for brain metastases.
* Participants who have received prophylactic cranial radiation for prevention of brain metastases
* Participants who cannot receive gadolinium
* Participants with stage IV-V chronic kidney disease or end stage renal disease
* Participants with widespread, definitive leptomeningeal disease
* Participants with a maximum tumor diameter exceeding 5 cm (if not resected)
* Participants with >6 definitive lesions consistent with brain metastases
* Participants with inadequate mental capacity to complete quality of life questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Death due to progressive neurologic disease | 12 months
  Clinical parameter to be assessed via review of study visits and medical records indicating cause of death (neurologic versus systemic)

SECONDARY OUTCOMES:
All-cause mortality | Until death or loss to follow up, up to 24 months
  Clinical parameter
Quality of life as assessed by patient Questionnaire | Until death or loss to follow up, up to 24 months
  Questionnaire - MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT)
Neurocognitive function: Verbal learning and memory | 12 months
  Hopkins Verbal Learning Test -Revised (HVLT-R)
Neurocognitive function: Visual attention and task switching | 12 months
  Trail Making Test Part A and B (TMT)
Neurocognitive function: Verbal fluency | 12 months
  Controlled Oral Word Association Test (COWAT)
Neurocognitive function: Cognitive impairment | 12 months
  Mini Mental Status Examination (MMSE)
Ability to complete activities of daily living | Until death or loss to follow up, up to 24 months
  Questionnaire - EQ-5D
Performance status | Until death or loss to follow up, up to 24 months
  Karnofsky performance status
Incidence and time to detection of new brain metastases | Until death or loss to follow up, up to 24 months
  Radiographic assessment of first appearance of new brain metastases
Incidence and time to local recurrence of existing brain metastases | Until death or loss to follow up, up to 24 months
  Radiographic assessment of first local recurrence in the 1-6 brain metastases that were initially treated with radiation
Incidence and time to development of radiation necrosis | Until death or loss to follow up, up to 24 months
  Radiographic assessment of first appearance of radiation necrosis
Incidence and time to development of leptomeningeal disease | Until death or loss to follow up, up to 24 months
  Radiographic assessment of first appearance of leptomeningeal disease
Incidence and time to progressive intracranial disease | Until death or loss to follow up, up to 24 months
  Radiographic assessment of first appearance of progressive intracranial disease
Incidence and time to salvage craniotomy | Until death or loss to follow up, up to 24 months
  Clinical assessment of first use of neurosurgical resection as salvage therapy
Incidence and time to additional CNS-directed radiotherapeutic treatments (stereotactic or WBRT) after the initial course | Until death or loss to follow up, up to 24 months
  Clinical assessment of first use of salvage brain-directed radiation
Incidence and time to the development of seizures | Until death or loss to follow up, up to 24 months
  Clinical assessment of first post-treatment seizure as assessed during routine study visits and via medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Ayal A Aizer, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aizer AA, Tanguturi SK, Shi DD, Catalano PJ, Shin KY, Ricca I, Johnson M, Benham G, Kozono DE, Mak RH, Hertan L, Chipidza F, Krishnan M, Pashtan I, Peng L, Qian JM, Shiloh RY, Cagney DN, Sands J, Brown PD, Wen PY, Haas-Kogan DA, Rahman R. Stereotactic Radiosurgery in Patients With Small Cell Lung Cancer and 1-10 Brain Metastases: A Multi-Institutional, Phase II, Prospective Clinical Trial. J Clin Oncol. 2025 Sep 20;43(27):2986-2997. doi: 10.1200/JCO-25-00056. Epub 2025 Jul 11. PMID 40644657